CLINICAL TRIAL: NCT06143670
Title: A Randomized, Controlled, Examiner-Blind Clinical Study Investigating the Effects of a Dentifrice Containing 0.454% w/w Stannous Fluoride on Gingivitis Treatment and Plaque Reduction When Used Twice Daily for 12 Weeks
Brief Title: A Clinical Study Investigating the Effects of a Dentifrice Containing 0.454% Stannous Fluoride on Gingivitis Treatment and Plaque Reduction When Used Twice Daily for 12 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300107
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): Participants will be instructed to brush their teeth with full ribbon of toothpaste (0.454% w/w SnF2) on head of toothbrush provided for at least one (timed) minute twice a day (morning and evening) for 12 weeks.
  Interventions: Drug: Stannous fluoride toothpaste
- Negative Control (Active Comparator): Participants will be instructed to brush their teeth with full ribbon of toothpaste (0.243% w/w Sodium fluoride) on head of toothbrush provided for at least one (timed) minute twice a day (morning and evening) for 12 weeks.
  Interventions: Drug: Sodium fluoride toothpaste

INTERVENTIONS:
Drug: Stannous fluoride toothpaste — 0.454% w/w SnF2
  Arms: Test Product
Drug: Sodium fluoride toothpaste — 0.243% w/w Sodium fluoride
  Arms: Negative Control

SUMMARY:
The purpose of this clinical study is to investigate the efficacy of a dentifrice containing 0.454 percent (%) weight by weight (w/w) stannous fluoride (SnF2), on gingivitis treatment and plaque reduction, compared to a regular fluoride dentifrice after 12 weeks twice daily brushing in a population of clinically diagnosed gingivitis without undergoing dental prophylaxis.

DETAILED DESCRIPTION:
This will be a single center, randomized, controlled, single blind (examiner blind), two-treatment arm, parallel study. Study participants will be over 18 years old, non-smokers, in good general health with clinically measurable levels of gingivitis that meet all study criteria at the Screening and Baseline visits. Approximately 160 participants (approximately 80 per group) will be randomized to ensure approximately 144 evaluable participants (approximately 72 per group) complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is at least 18 years old, inclusive.
* A participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant/relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the participant's ability to understand and follow study procedures and requirements.
* Participant oral health that meets all the following:

At Screening (Visit 1):

1. Participant with at least 20 natural, permanent teeth.
2. Participant with at least 40 evaluable surfaces for MGI, BI, and TPI (An evaluable surface is defined as having two thirds of the natural tooth surface gradable for the selected clinical indices. The following will not be included in the evaluable surface count: third molars; fully crowned/extensively restored, grossly carious, orthodontically banded/bonded or abutment teeth; surfaces with calculus deposits which, in the opinion of the clinical examiner, would interfere with the baseline assessments of the selected clinical indices).
3. A participant with plaque-induced gingivitis, in the opinion of the clinical examiner, as confirmed by a gross visual examination.

   At Baseline (Visit 2):
4. A participant with ongoing hard tissue eligibility and, in the opinion of the clinical examiner, at least 40 evaluable surfaces.
5. A participant with 10% to 30% bleeding sites (following BI).
6. A participant with mean whole mouth TPI score >=1.5.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a sponsor's employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who has any other clinical serious or unstable conditions (for example, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) which could have affected study outcomes and/or participant safety.
* A participant who is a pregnant female (self-reported) or is intending to become pregnant over the duration of the study.
* A participant who is a breastfeeding female.
* A participant who is known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who is unwilling or unable to comply with the lifestyle considerations.
* Participant who is a current smoker or an ex-smoker who stopped within 6 months of Screening.
* Participant who is using smokeless forms of tobacco (for example, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed xerostomia or is taking any medication that in the view of the investigator is causing xerostomia.
* A participant who has a medical condition which could have directly influenced gingival bleeding (for example, type 2 diabetes).
* A participant who has a bleeding disorder that could have affected study outcomes and/or participant safety.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (for example, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.
* Medication exclusions at screening (Visit 1):

  1. A participant using any antibiotic medication within 14 days prior to screening or at any time during the study.
  2. A participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
  3. A participant currently taking a systemic medication (for example, anti-inflammatory, anticoagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (for example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
* Medication exclusions at Baseline (Visit 2):

  1. A participant who has taken (in the previous 14 days), any antibiotics.
  2. A participant who has taken (in the previous 14 days) a systemic medication (for example, anti-inflammatory, anti-coagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (for example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
  3. A participant who has used an antibacterial dentifrice or mouthwash (for example, chlorhexidine) or any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, in the period between Screening and the Baseline visit.
* Periodontal exclusions:

  1. A participant who shows signs of active periodontitis (with probing pocket depths greater than [>] 3mm).
  2. A participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
  3. A participant who has gingivitis, which in the opinion of the investigator, is not expected to respond to treatment with an over the counter (OTC) dentifrice.
* Dental Exclusions:

  1. A participant who has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  2. A participant who has dentures (partial or full).
  3. A participant who has an orthodontic appliance (bands, appliances, or fixed/ removable retainers).
  4. A participant who received orthodontic therapy within 3 months of Screening.
  5. A participant who has numerous restorations in a poor state of repair.
  6. A participant who has any dental condition (for example, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  7. A participant who has had dental prophylaxis within 12 weeks of Screening.
  8. A participant who has had teeth bleaching within 12 weeks of Screening.
  9. A participant who has high levels of extrinsic stain or calculus deposits, in the opinion of the investigator, that could have interfered with plaque assessments.
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 162 participants were screened of which 159 participants were enrolled, and 152 participants were randomized to receive treatment in 2 groups: Test Product group (76 participants) and Reference Product group (76 participants). 10 participants were not randomized (7 participants did not meet the study criteria, 2 participants withdrew consent, and 1 participant had an adverse event [AE]). A total of 148 randomized participants completed the study.
Groups:
- Test Product: Participants were instructed to apply a ribbon of test toothpaste (Parodontax Complete Protection) containing 0.454 percent (%) weight by weight (w/w) stannous fluoride (SnF2) across the full brush head of toothbrush provided and brush their teeth for at least one (timed) minute twice daily (morning and evening) for 12 weeks.
- Reference Product (Negative Control): Participants were instructed to apply a ribbon of reference toothpaste (Crest Cavity Protection) containing 0.243% w/w sodium fluoride across the full brush head of toothbrush provided and brush their teeth for at least one (timed) minute twice daily (morning and evening) for 12 weeks.
Period: Overall Study
Arm/Group | Test Product | Reference Product (Negative Control)
Started | 76 | 76
Completed | 73 | 75
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received at least one dose of the study product.
Groups:
- Test Product: Participants were instructed to apply a ribbon of test toothpaste (Parodontax Complete Protection) containing 0.454% w/w SnF2 across the full brush head of toothbrush provided and brush their teeth for at least one (timed) minute twice daily (morning and evening) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product (Negative Control) | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (14.00) | 50.5 (13.04) | 49.2 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 119
  Male | 17 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 73 | 73 | 146
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 8 | 9 | 17
  American Indian or Alaskan Native | 1 | 0 | 1
  White - Arabic/North African Heritage | 2 | 0 | 2
  White - White/Caucasian/European Heritage | 64 | 65 | 129
  Multiple | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in the Number of Bleeding Sites (NBS) at Week 12
Description: The NBS were calculated using the bleeding index (BI) assessment. BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. The BI was assessed on the facial and lingual gingival surfaces of each scorable tooth using PCP11.5B Hu-Friedy Qulix Color Coded probe. The probe was gently inserted into the gingival crevice to a depth of approximately 1 millimeter (mm) and then run around the tooth gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. NBS for each participant was calculated as the number of evaluable tooth sites with bleeding observed immediately on probing or within 30 seconds of probing. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 12. Baseline was defined as Day 0. A negative change from Baseline indicated improvement in gingival condition.
Time Frame: Baseline and Week 12
Population: Modified Intent-To-Treat (mITT) population included all randomized participants who completed at least one use of study product and had at least one post baseline clinical performance assessment.
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Product
Number analyzed (Participants) | 73
bleeding sites | -14.6 (0.99)
Statistical Analysis 1: Comparison: Test Product; Change from Baseline at Week 12 (Test for non-zero within group change from Baseline); Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

2. Secondary Outcome: Adjusted Mean Change From Baseline in the NBS at Week 12 (Test Product Versus [vs.] Reference Product)
Description: The NBS were calculated using the BI assessment. BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. The BI was assessed on the facial and lingual gingival surfaces of each scorable tooth using PCP11.5B Hu-Friedy Qulix Color Coded probe. The probe was gently inserted into the gingival crevice to a depth of approximately 1 mm and then run around the tooth gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. NBS for each participant was calculated as the number of evaluable tooth sites with bleeding observed immediately on probing or within 30 seconds of probing. Change from Baseline was calculated by subtracting the Baseline value from the value at Week 12. Baseline was defined as Day 0. A negative change from Baseline indicated improvement in gingival condition.
Time Frame: Baseline and Week 12
Population: mITT population. Here, overall number analyzed is defined as the number of participants with data available for analysis of this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Product | Reference Product (Negative Control)
Number analyzed (Participants) | 73 | 75
bleeding sites | -14.6 (0.99) | 2.2 (0.98)
Statistical Analysis 1: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -16.9, 95% CI 2-sided [-19.6 to -14.1], Standard Error of Mean 1.40 — Adjusted mean difference was calculated as test product minus reference product

3. Secondary Outcome: Adjusted Mean Change From Baseline in the NBS at Week 3 and Week 6 (Test Product vs. Reference Product)
Description: The NBS were calculated using the BI assessment. BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. The BI was assessed on the facial and lingual gingival surfaces of each scorable tooth using PCP11.5B Hu-Friedy Qulix Color Coded probe. The probe was gently inserted into the gingival crevice to a depth of approximately 1 mm and then run around the tooth gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. NBS for each participant was calculated as the number of evaluable tooth sites with bleeding observed immediately on probing or within 30 seconds of probing. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. Baseline was defined as Day 0. A negative change from Baseline indicated improvement in gingival condition.
Time Frame: Baseline, Week 3 and Week 6
Population: mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: bleeding sites
Arm/Group | Test Product | Reference Product (Negative Control)
Number analyzed (Participants) | 73 | 76
bleeding sites
  Change from Baseline at Week 3: number analyzed (Participants) | 70 | 75
  Change from Baseline at Week 3 | -14.8 (1.05) | 1.2 (1.01)
  Change from Baseline at Week 6: number analyzed (Participants) | 72 | 76
  Change from Baseline at Week 6 | -16.7 (0.84) | 0.9 (0.82)
Statistical Analysis 1: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 3; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -16.0, 95% CI 2-sided [-18.9 to -13.1], Standard Error of Mean 1.46 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 6; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -17.6, 95% CI 2-sided [-19.9 to -15.3], Standard Error of Mean 1.17 — Adjusted mean difference was calculated as test product minus reference product

4. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Overall Turesky Plaque Index (TPI) at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: TPI was used to assess plaque on the facial and lingual surfaces of each scorable tooth. The plaque was first disclosed using a plaque disclosing dye solution, disclosed plaque was then scored on a 6-point scale ranging from 0 to 5, where 0=No plaque; 1=Separate flecks of plaque at the cervical margin; 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin; 3=Band of plaque wider than 1 mm but covering less than one third of the tooth surface; 4=Plaque covering more than one third but less than two thirds of the tooth surface; 5=Plaque covering more than two thirds of the tooth surface. Overall TPI score for each participant=Sum of index values over all evaluable tooth sites (sites scored as 0 to 5), divided by the number of evaluable tooth sites and ranged from 0 to 5. Lower score=better outcome. Change from Baseline=Value at each indicated timepoint minus Baseline value. Baseline=Day 0. A negative change from Baseline indicated improvement (less plaque accumulation).
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product | Reference Product (Negative Control)
Number analyzed (Participants) | 73 | 76
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 70 | 75
  Change from Baseline at Week 3 | -0.30 (0.026) | -0.02 (0.025)
  Change from Baseline at Week 6: number analyzed (Participants) | 72 | 76
  Change from Baseline at Week 6 | -0.29 (0.023) | -0.10 (0.023)
  Change from Baseline at Week 12: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 12 | -0.32 (0.025) | -0.03 (0.024)
Statistical Analysis 1: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 3; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.28, 95% CI 2-sided [-0.35 to -0.20], Standard Error of Mean 0.036 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 6; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.20, 95% CI 2-sided [-0.26 to -0.13], Standard Error of Mean 0.032 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.29, 95% CI 2-sided [-0.36 to -0.22], Standard Error of Mean 0.035 — Adjusted mean difference was calculated as test product minus reference product

5. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Interproximal TPI at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: TPI was used to assess plaque on the facial and lingual surfaces of each scorable tooth. The plaque was first disclosed using a plaque disclosing dye solution and scored on a 6-point scale ranging from 0 to 5, where 0=No plaque; 1=Separate flecks of plaque at the cervical margin; 2=Thin continuous band of plaque (up to 1 mm) at the cervical margin; 3=Band of plaque wider than 1 mm but covering less than one third of the tooth surface; 4=Plaque covering more than one third but less than two thirds of the tooth surface; 5=Plaque covering more than two thirds of the tooth surface. Interproximal TPI score for each participant=Sum of index values over all evaluable distal and mesial tooth sites, divided by the number of evaluable distal and mesial tooth sites and ranged from 0 to 5. Lower score=better outcome. Change from Baseline=Value at each indicated timepoint minus Baseline value. Baseline=Day 0. A negative change from Baseline indicated improvement (less plaque accumulation).
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product | Reference Product (Negative Control)
Number analyzed (Participants) | 73 | 76
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 70 | 75
  Change from Baseline at Week 3 | -0.23 (0.022) | -0.02 (0.021)
  Change from Baseline at Week 6: number analyzed (Participants) | 72 | 76
  Change from Baseline at Week 6 | -0.25 (0.020) | -0.09 (0.019)
  Change from Baseline at Week 12: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 12 | -0.28 (0.022) | -0.04 (0.021)
Statistical Analysis 1: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 3; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.22, 95% CI 2-sided [-0.28 to -0.16], Standard Error of Mean 0.030 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 6; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.16, 95% CI 2-sided [-0.21 to -0.10], Standard Error of Mean 0.028 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.24, 95% CI 2-sided [-0.30 to -0.18], Standard Error of Mean 0.030 — Adjusted mean difference was calculated as test product minus reference product

6. Secondary Outcome: Adjusted Mean Change From Baseline in BI at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: BI assesses the number of bleeding points elicited on probing as a measure of gingival condition. BI was assessed on the facial and lingual gingival surfaces of each scorable tooth using PCP11.5B Hu-Friedy Qulix Color Coded probe. Gingival bleeding was scored on a 3-points scale with scores ranging from 0 to 2, where 0=No bleeding after 30 seconds, 1=Bleeding observed within 30 seconds of probing, 2=Bleeding observed immediately on probing. BI score for each participant=sum of index values over all evaluable tooth sites (those scored as 0, 1, or 2), divided by the number of evaluable tooth sites. Lower score=better outcome. Change from Baseline was calculated by subtracting the Baseline value from the value at each indicated timepoint. Baseline=Day 0. A negative change from Baseline indicated improvement in gingival condition.
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product | Reference Product (Negative Control)
Number analyzed (Participants) | 73 | 76
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 70 | 75
  Change from Baseline at Week 3 | -0.12 (0.009) | 0.01 (0.009)
  Change from Baseline at Week 6: number analyzed (Participants) | 72 | 76
  Change from Baseline at Week 6 | -0.14 (0.007) | 0.01 (0.007)
  Change from Baseline at Week 12: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 12 | -0.12 (0.009) | 0.01 (0.009)
Statistical Analysis 1: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 3; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.12, 95% CI 2-sided [-0.15 to -0.10], Standard Error of Mean 0.013 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 6; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.15, 95% CI 2-sided [-0.17 to -0.13], Standard Error of Mean 0.010 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.14, 95% CI 2-sided [-0.16 to -0.11], Standard Error of Mean 0.013 — Adjusted mean difference was calculated as test product minus reference product

7. Secondary Outcome: Adjusted Mean Change From Baseline in Modified Gingival Index (MGI) at Weeks 3, 6 and 12 (Test Product vs. Reference Product)
Description: MGI assessment is a non-invasive evaluation which focuses on visual symptoms of gingivitis (example, redness, texture, edema). MGI was assessed on facial and lingual surfaces of each scorable tooth and scored on a 5-point scale ranging from 0 to 4, where 0=Absence of inflammation; 1=Mild inflammation; slight change in color, little change in color; little change in texture of any portion of marginal or papillary gingival unit; 2=Mild inflammation; criteria as 1 but involving entire marginal or papillary gingival unit; 3=Moderate inflammation; glazing, redness, edema, and/or hypertrophy of marginal or papillary gingival unit; 4=Severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicated better outcome. Change from Baseline=Value at each indicated timepoint minus Baseline [Day 0] value. A negative change from Baseline indicated improvement in symptoms.
Time Frame: Baseline, Weeks 3, 6 and 12
Population: mITT Population. Only those participants available at the indicated timepoints were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Test Product | Reference Product (Negative Control)
Number analyzed (Participants) | 73 | 76
score on a scale
  Change from Baseline at Week 3: number analyzed (Participants) | 70 | 75
  Change from Baseline at Week 3 | -0.51 (0.037) | 0.12 (0.036)
  Change from Baseline at Week 6: number analyzed (Participants) | 72 | 76
  Change from Baseline at Week 6 | -0.71 (0.032) | -0.07 (0.032)
  Change from Baseline at Week 12: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 12 | -0.71 (0.034) | -0.03 (0.034)
Statistical Analysis 1: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 3; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.64, 95% CI 2-sided [-0.74 to -0.53], Standard Error of Mean 0.052 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 2: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 6; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.65, 95% CI 2-sided [-0.74 to -0.56], Standard Error of Mean 0.045 — Adjusted mean difference was calculated as test product minus reference product
Statistical Analysis 3: Comparison: Test Product vs Reference Product (Negative Control); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures; Adjusted Mean Difference = -0.67, 95% CI 2-sided [-0.77 to -0.58], Standard Error of Mean 0.048 — Adjusted mean difference was calculated as test product minus reference product

ADVERSE EVENTS:
Time Frame: From signing of informed consent form until 5 days after last administration of study product or last study procedure (up to approximately 111 days).
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) was a particular category of an AE where the adverse outcome is serious.
Arm/Group | Test Product | Reference Product (Negative Control)
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 5/76 | 7/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product (N=76) | Reference Product (Negative Control) (N=76)
ORAL MUCOSAL EXFOLIATION (Gastrointestinal disorders) | 4 | 2
APHTHOUS ULCER (Gastrointestinal disorders) | 1 | 2
HYPERAESTHESIA TEETH (Gastrointestinal disorders) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
MOUTH INJURY (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT06143670/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT06143670/SAP_001.pdf